CLINICAL TRIAL: NCT03054974
Title: Traditional Chinese Medicine Clinical Practice Rehabilitation of Post-stroke Spasticity
Brief Title: TCM Clinical Practice Rehabilitation of Post-stroke Spasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, JiangFeng, JiangFeng Clinical Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013BAI10B04
Record Dates: First submitted 2016-11-20; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Stroke
Keywords: Stroke; Traditional Chinese Medicine; Rehabilitation
MeSH Terms: conditions — Stroke | interventions — Medicine, Tibetan Traditional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Modern rehabilitation treatment (Experimental): Modern rehabilitation treatment
  Interventions: Other: Modern rehabilitation treatment
- Modern rehabilitation &TCM (Experimental): Modern rehabilitation treatment and traditional Chinese medicine
  Interventions: Other: Modern rehabilitation &TCM
- modern rehabilitation &Baimai Ruangao (Experimental): modern rehabilitation treatment and Baimai Ruangao
  Interventions: Other: modern rehabilitation &Baimai Ruangao
- modern rehabilitation &Tibetan medicine (Experimental): modern rehabilitation treatment and Tibetan medicine treatment
  Interventions: Other: modern rehabilitation &Tibetan medicine

INTERVENTIONS:
Other: Modern rehabilitation treatment — PT 1 hour per day and OT 30min per day
  Arms: Modern rehabilitation treatment
Other: Modern rehabilitation &TCM — Traditional Chinese Medicine, including massage and medicated bath
  Arms: Modern rehabilitation &TCM
Other: modern rehabilitation &Baimai Ruangao — modern rehabilitation treatment with Baimai Ruangao and massage
  Arms: modern rehabilitation &Baimai Ruangao
Other: modern rehabilitation &Tibetan medicine — modern rehabilitation treatment and Tibetan medicine(medicated bath with wuweiganlu and rub with baimairuangao)
  Arms: modern rehabilitation &Tibetan medicine

SUMMARY:
The purpose of this study is to determine the effectiveness,safety and Input-output ratio of chinese traditional treatment in spasm after stroke,both in massage and herbal medicine bathing.

DETAILED DESCRIPTION:
A Muti-center randomized controlled study with large samples to observe improvement of motor function,severity of spasm,ADL(activity of daily lives),by standardized protocols of TCM techniques(massage and herbal bathing) combined with conventional rehabilitation on spasm after stroke in 1 month.Modified Ashworth scale,Fugl-Meyer Index and Modified barthel Index were used for spasm,motor function and ADL.And also the follow up research within 3 months and 6 months focus on the efficacy duration of TCM on spasm.Try to find suitable timing for intervention on spasm by CTM(Massage and herbal medicine bathing)and the connection between spasm severity and treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria of stroke and diagnosed by CT or MRI
* Patient must be between the ages of 18 and 85 years.
* All patients were examined at least 1 month after stroke and less than 12 months.
* At least a set of spasmous muscles' level ≥1+ of dysfunctional extremities (modified Ashworth scale)
* Body movement function decreased significantly.
* The doses and kinds of anticonvulsant drugs should be used stable for more than 1 month if they are used
* Patient must understand and be willing, able and likely to comply with all study procedures.
* Patient must be able to give voluntary written informed consent.

Exclusion Criteria:

* Significant cognitive defects(MMSE<16)，unable to finish the Fugl-Meyer scale,etc..
* Other significant limb diseases such as fracture, severe arthritis,amputation
* Joint contracture formation
* Patients with significant pain and swelling suffering from complex regional syndrome after acute stroke
* Accept botulinum toxin or alcohol nerve block 3 months prior to the start of the experiment
* Patients need nerve block at any point of time during the whole experiment procedure.
* Serious cardiac,hepatic or renal insufficiency and patients with shock.
* Limb skin of patients who need medicated is visible wound.
* Patients with cancer or pregnancy
* Patients who participate in other clinical studies within 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1208 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 6 months
  the common used clinical measurement to assess the levels of limb spasticity

SECONDARY OUTCOMES:
Fugl-Meyer Moter Assessment | 6 months

OTHER OUTCOMES:
Barthel Index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Li jianan, Doctor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No